CLINICAL TRIAL: NCT02588222
Title: GRINCH: Groningen Initiative on Reference Intervals in Children
Acronym: GRINCH
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Cisbio Bioassays (Industry)
Responsible Party: Principal Investigator, P.F. van Rheenen, Dr., University Medical Center Groningen
Other Study IDs: 201500284
Record Dates: First submitted 2015-08-07; First posted 2015-10-27 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — feces samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy children: Healthy children, aged 6-18 years old.

SUMMARY:
The purpose of this study is to establish reliable reference intervals for fecal S100A12 in healthy children.

DETAILED DESCRIPTION:
RATIONALE S100A12 (calgranulin C) is a cytoplasmic protein secreted exclusively by activated neutrophils. It can be measured in stools and elevated levels are observed in children with inflammatory bowel disease. The protein is stable in stool samples for up to seven days at room temperature, which allows collection at home and potential delays in transport to the laboratory. S100A12 could be used as a marker to discriminate between pediatric inflammatory and functional gastro-intestinal conditions, and prevent children with a low probability of inflammation from unnecessary endoscopic procedures. Until now a reliable reference interval for healthy children is lacking.

OBJECTIVE To establish reliable reference intervals for fecal S100A12 in healthy children.

TIME FRAME Healthy children will be asked to send in one feces sample anonymously during the inclusion period. The investigators expect that the required 120 samples will be collected before December 2015. There will be no follow up of patients.

ELIGIBILITY:
Inclusion Criteria healthy volunteers:

* Age: 6-18 years old

Exclusion Criteria:

* Treated for any gastro-intestinal symptoms
* Diarrhea in the last week before the collection of the feces sample
* Fever in the last week before collection of the feces sample
* Use of NSAIDs of Proton pump inhibitors in the last 14 days before collection feces sample.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy children, aged 6-18 years old
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Levels of Calgranulin C (S100A12) in healthy children | One measurement at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Patrick van Rheenen, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands